CLINICAL TRIAL: NCT00848705
Title: Adolescent Self-Management of Type 1 Diabetes: an Intervention
Brief Title: Adolescent Self-Management of Type 1 Diabetes: an Intervention (Completed)
Acronym: YourWay
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Shelagh Mulvaney, PhD, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DK70026-01A2
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2011-01

CONDITIONS: Adolescent Type 1 Diabetes
Keywords: type 1 diabetes, adolescent, self-management
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Measurement Only (Active Comparator)
  Interventions: Behavioral: YourWay Internet Intervention
- Internet Intervention (Experimental)
  Interventions: Behavioral: YourWay Internet Intervention

INTERVENTIONS:
Behavioral: YourWay Internet Intervention — The intervention is an 11 week program that teaches problem solving of barriers to self-management.

SUMMARY:
The goals of this R21 exploratory pilot and feasibility study were to: 1) design an Internet-based self-management intervention for adolescents with type 1 diabetes; 2) test that intervention in a small randomized trial to establish technical feasibility, intervention acceptability, and competence in completing the necessary recruitment and research procedures. Although not powered to detect statistically significant changes, possible outcomes of this study include improvements in problem-solving, coping, and self-management behaviors.

ELIGIBILITY:
Inclusion Criteria:diagnosed for at least 6 months, age 13-17; Internet access, parental consent -

Exclusion Criteria: Any sensory deficits that would preclude seeing or hearing.

-

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2007-10; Primary Completion 2009-01 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Self-management behaviors | End of intervention

SECONDARY OUTCOMES:
Self-management Problem solving | end of study period

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States